CLINICAL TRIAL: NCT01219608
Title: Iranian Intensive Care Unit (ICU) Glutamine Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr Reza Rastmanesh, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: eums1388
Record Dates: First submitted 2010-10-06; First posted 2010-10-13 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2010-10

CONDITIONS: Trauma Patients in ICU
MeSH Terms: interventions — Glutamine; Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glutamine 0.5 g/kg/day (Active Comparator)
  Interventions: Dietary Supplement: Glutamine 0.5 g/kg/day
- Glutamine 1 g/kg/day (Active Comparator)
  Interventions: Dietary Supplement: Glutamine 1 g/kg/day
- Enteral Nutrition (Placebo Comparator)
  Interventions: Dietary Supplement: Enteral Nutrition

INTERVENTIONS:
Dietary Supplement: Glutamine 0.5 g/kg/day — Glutamine 0.5 g/kg/day
  Arms: Glutamine 0.5 g/kg/day
Dietary Supplement: Glutamine 1 g/kg/day — Glutamine 1 g/kg/day
  Arms: Glutamine 1 g/kg/day
Dietary Supplement: Enteral Nutrition — Ordinary Enteral Nutrition
  Arms: Enteral Nutrition

SUMMARY:
This is a double-blinded placebo-controlled block randomized study in intensive care patients comparing enteral glutamine supplementation to placebo. The hypothesis is an improvement of clinical and paraclinical outcomes. The primary endpoint is Infection Probability Score (IPS) and Systemic Inflammatory Response Syndrome (SIRS). Anthropometric measures and serum inflammatory mediators will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* No corticosteroids use
* No history of heart, liver and kidney diseases
* Nutrition through nasogastric or orogastric

Exclusion Criteria:

* Patients who will not tolerate enteral nutrition for more than 48 hours
* Patients who are NPO and nutritional support has not started
* Lactating and pregnant women
* Kidney failure during the study
* A history of glutamin supplement use before the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Infection Probability Score | 10 days after intervention
  Infection Probability Score will be measured and will be compared to the baseline after 10 days of the intervention
Systemic Inflammatory Response Syndrome | 10 days after intervention
  Systemic Inflammatory Response Syndrome will be measured and will be compared to the baseline after 10 days of the intervention

SECONDARY OUTCOMES:
Prealbumin | 10 days after intervention
  Prealbumin will be measured and will be compared to the baseline after 10 days of the intervention
CRP | 10 days after intervention
  CRP will be measured and will be compared to the baseline after 10 days of the intervention
Serum prealbumin | 10 days after the intervention
  Prealbumin will be measured and will be compared to the baseline after 10 days of the intervention
Length of stay (LOS)
  LOS will be measured and will be compared to the baseline after 10 days of the intervention
Bed sores | 10 days after intervention
  Bed sores will be measured and will be compared to the baseline after 10 days of the intervention
Mechanical ventilation | 10 days after intervention
  Mean mechanical ventilation need will be measured and will be compared to the baseline after 10 days of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahra Hospital, Isfahan, Isfahan, Iran